CLINICAL TRIAL: NCT06718894
Title: Multitarget Strategy for Primary Podocytopathies
Acronym: PODO-TARGET
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Collaborators: Fondazione Regionale per la Ricerca Biomedica (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 5387
Record Dates: First submitted 2024-12-02; First posted 2024-12-05 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-11

CONDITIONS: Nephrotic Syndrome
Keywords: podocytopathy; transplant
MeSH Terms: conditions — Nephrotic Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Biologic fluid sampling — The only interventions in addition to standard clinical practice will be blood sampling, the collection of morning spot urine and the collection of the discarded effluent of the plasmapheresis procedure (when performed according to clinical indication).

SUMMARY:
The goal of this clinical trial is to verify whether a cell culture system can be used to evaluate the presence of a factor capable of causing proteinuria in the serum of patients with primary podocytopathies. This system will also be used to evaluate the in vitro efficacy of a combined therapy for the treatment of this disorder.

Researchers will compare samples from patients with primary podocytopathies with those obtained from healthy subjects and patients with other renal disorders.

Participants will be asked to visit the clinic at regular intervals for up to 36 months, and to provide blood and urine samples (and a sample of the discarded plasmapheresis effluent in case the procedure is performed).

ELIGIBILITY:
Inclusion Criteria:

* Signature of informed consent for study participation
* One of the following conditions:

  1. Patients with primary podocytopathies (with a histological diagnosis of FSGS or MCD) showing clinical and/or histological evidence of post-transplant recurrence.
  2. Patients with primary podocytopathies (with a histological diagnosis of FSGS or MCD) without clinical and/or histological evidence of post-transplant recurrence.
  3. Patients with primary podocytopathies in their native kidneys in an active clinical phase of the disease.
  4. Patients with podocytopathies presenting clinical features compatible with a secondary form due to another condition.
  5. Patients with glomerulonephritis other than primary podocytopathies (e.g., IgA nephropathy, systemic lupus erythematosus, membranous nephropathy).
  6. Patients with no history of renal diseases

Exclusion Criteria:

* Subjects affected by primary podocytopathies or other glomerulonephritides in clinical remission or with ESRD (eGFR < 15 ml/min) and/or on renal replacement therapy
* Individuals unable to understand and consent to the study procedures
* Any clinical condition that, according to the investigator's judgment, could compromise patient safety during study participation

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-12 (Estimated); Primary Completion 2032-01 (Estimated); Study Completion 2032-11 (Estimated)

PRIMARY OUTCOMES:
Co-culture system capability to distinguish recurrent podocytopathies from healthy subjects | Baseline
  The difference in the increase of albumin permeability in the endothelium-podocyte co-culture system after exposure to serum from patients with recurrent podocytopathies and healthy subjects will be compared.

SECONDARY OUTCOMES:
In-vitro efficacy of SGLT2-inhibitors and uPAR/FPR-inhibitors on primary podocytopathies | Baseline, 16 weeks and in case of remission/recurrence
Co-culture system capability to distinguish recurrent podocytopathies from other glomerular disorders | Baseline
  The difference in the increase of albumin permeability in the endothelium-podocyte co-culture system after exposure to serum from patients with recurrent podocytopathies and patients with other glomerular disorders will be compared.
Co-culture system reliability in case of podocytopathy remission | Baseline, 16 weeks and in case of remission/recurrence
  The difference in the increase of albumin permeability in the endothelium-podocyte co-culture system after exposure to serum from patients with active podocytopathies and podocytopathies in the remission phase will be compared.

OTHER OUTCOMES:
Podocytopathy-specific proteomic and metabolomic profile in serum/plasma and urine | Baseline, 16 weeks and in case of remission/recurrence
Podocytopathy-specific proteomic and metabolomic profile of endothelial cells and podocytes exposed to serum from patients with podocytopathies | Baseline, 16 weeks and in case of remission/recurrence
Podocytopathy-specific in vitro activation of immune subsets | Baseline, 16 weeks and in case of remission/recurrence
Podocytopathy-specific transcriptomic signatures of different immune cell subsets | Baseline, 16 weeks and in case of remission/recurrence
Podocytopathy-specific genomic differences in variants and SNPs associated with increased risk of disease | Baseline
Podocytopathy-specific proteomic and transcriptomic profile in kidney tissue | Baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided